CLINICAL TRIAL: NCT00487071
Title: Efficacy of Anal Fistula Plug in the Management of High-type Anal Fistulae: a Pilot Study
Brief Title: Anal Fistula Plug for High-type Anal Fistulae
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No financial support
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon S. M. Ng, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2006.274
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: High-type Anal Fistulae
Keywords: Anal fistula; High-type; Anal fistula plug; Efficacy; Recurrence
MeSH Terms: conditions — Rectal Fistula; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anal fistula plug (Experimental)
  Interventions: Device: Anal fistula plug

INTERVENTIONS:
Device: Anal fistula plug

SUMMARY:
The aim of this pilot study is to evaluate the efficacy and safety of anal fistula plug in the management of high-type anal fistulae among Hong Kong Chinese patients.

DETAILED DESCRIPTION:
An anal fistula is an abnormal communication between the anal or rectal lumen and the perianal skin. Anal fistulae are described according to the level at which they transgress the anal sphincter. If the internal opening begins above the anal sphincter then the fistula is described as 'high'. Traditional surgery for high-type anal fistulae often requires staged operations with fistulotomy and seton insertion. The surgery usually results in large and deep wounds which can take months to heal. Moreover, risk of faecal incontinence is inevitable because part of the anal sphincter is divided during the surgery.

The Surgisis® anal fistula plug is a minimally invasive and sphincter-preserving alternative to traditional fistula surgery. It is a newly developed biomaterial made from complex collagen obtained from pigs - animals that have a collagen structure almost identical to that of human tissue. During manufacturing of the plug, living cells are removed by special processes to help ensure that no transmittable diseases are present in the tissue. The plug is a conical device and is placed by drawing it through the fistula tract and suturing it in place. As pig collagen is so similar to human collagen, the plug, once implanted, incorporates naturally over time into the human tissue (human cells and tissues will 'grow' into the plug), thus facilitating the closure of the fistula. Preliminary clinical data from USA showed a high fistula closure rate of 87%. The anal fistula plug can also avoid protracted postoperative wound care and minimise the risk of faecal incontinence.

We would like to carry out a pilot study, the aim of which is to evaluate the efficacy and safety of this new anal fistula plug in the management of high-type anal fistulae. This is believed to be the first study of its kind in Hong Kong.

Patients with high-type anal fistulae confirmed by MRI will be recruited into this study. Patients with previous history of fistula surgery, patients with Crohn's disease, and patients with known allergy to porcine material will be excluded. EUA + anal fistula plug will be performed. Outcome measures include fistula healing rate, recurrence rate, and morbidity. Follow-up MRI will be arranged at 3 months and 6 months after the operation to objectively evaluate the healing of the fistulae.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high-type anal fistulae confirmed by MRI
* Informed consent available

Exclusion Criteria:

* Patients with previous fistula surgery
* Patients with Crohn's disease
* Patients allergic to porcine material

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Fistula healing rate and time for fistula closure | Up to 1 year

SECONDARY OUTCOMES:
Fistula recurrence rate | Up to 1 year
Morbidity | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Simon SM Ng, FRCSEd (Gen), Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Surgery, Prince of Wales Hospital, Hong Kong SAR, China